CLINICAL TRIAL: NCT07298239
Title: A Single-Center, Open-Label, Single-Arm, Exploratory Clinical Study to Evaluate the Safety and Efficacy of Allogeneic CAR-NK Cell Therapy in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Allogeneic CAR-NK Cell Therapy for Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XINGNIANZENG, Vice President of the Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25/216-0216
Record Dates: First submitted 2025-11-24; First posted 2025-12-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Biological: anti-PSMA CAR-NK

INTERVENTIONS:
Biological: anti-PSMA CAR-NK — Targeting PSMA CAR-NK cells

SUMMARY:
This study introduces a new treatment approach for metastatic castration-resistant prostate cancer, a stage of disease that remains difficult to manage with current therapies. Prostate cancer is the second most common cancer in men worldwide, and many patients eventually progress to an advanced, treatment-resistant stage despite hormone therapy, newer hormonal agents, or chemotherapy. Patients with metastatic castration-resistant disease often face a poor prognosis, complications such as bone metastases, and significant impacts on quality of life, highlighting the urgent need for new treatment options. This research focuses on an innovative immunotherapy using allogeneic anti-PSMA CAR-NK cells, which are engineered natural killer cells designed to precisely recognize and kill prostate cancer cells expressing the prostate-specific membrane antigen. CAR-NK cells combine the natural tumor-killing ability of NK cells with enhanced targeting and reduced immune escape, offering a potentially safer and more effective strategy. Through this clinical study, the safety, tolerability, and preliminary effectiveness of anti-PSMA CAR-NK cell therapy will be evaluated, aiming to provide new evidence and expand future treatment possibilities for patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male;
* Diagnosis of metastatic castration-resistant prostate cancer (mCRPC) meeting the following criteria: ① Serum testosterone at castration level: < 50 ng/dL or < 1.7 nmol/L; ② Meeting any one of the following conditions: a. PSA progression: Three consecutive rises in PSA measured at intervals of at least 1 week, with two increases being ≥ 50% above the PSA nadir, and a PSA value > 2 ng/mL; b. Radiographic progression: Two or more new lesions detected on bone scan, or an increase in soft tissue lesions assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST).
* Expected survival ≥ 6 months;
* ECOG performance status of 0-2;
* Positive prostate-specific membrane antigen (PSMA) expression;
* Voluntarily participate, provide written informed consent, and be able to comply with follow-up.

Exclusion Criteria:

* Prior treatment with other cell therapy products besides the investigational product, such as dendritic cells (DC), cytokine-induced killer cells (CIK), T cells, natural killer cells (NK), chimeric antigen receptor T-cell immunotherapy (CAR-T), etc.;
* History of other malignancies within 5 years prior to screening (except for completely resolved carcinoma in situ or malignancies deemed by the investigator to be slow-progressing);
* Abnormal function of major organs: a. Absolute neutrophil count (ANC) < 1.5 × 10⁹/L; Platelet count (Plt) < 100 × 10⁹/L; Hemoglobin (Hb) < 9 g/dL; b. Liver function: Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≥ 2.5 × the upper limit of normal (ULN) (or ≥ 5 × ULN for subjects with liver metastases); c. Renal function: Serum creatinine (Cr) ≥ 1.5 × ULN; d. Coagulation function: Prothrombin time (PT), Activated partial thromboplastin time (APTT), International Normalized Ratio (INR) ≥ 1.5 × ULN;
* Any currently treated active (viral, bacterial, fungal) infection, or any infection within the past 6 weeks requiring intravenous antibiotics for 7 days or longer, or any active infection requiring oral antibiotics within the past week;
* Active autoimmune disease, or history of severe autoimmune disease requiring long-term immunosuppressive therapy;
* Participation in another clinical trial study within 3 months;
* Inability to employ effective contraceptive measures;
* History of hypersensitivity to biologic macromolecular drugs;
* Untreated chronic active hepatitis B, or chronic hepatitis B virus carriers with HBV DNA ≥ 1000 copies/mL, or patients with active hepatitis C;
* Subjects deemed by the investigator to be unsuitable for participation in this study for other reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v5.0 | Baseline to 1 year post infusion
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
The pharmacokinetic analysis of Anti-PSMA CAR-NK Cell | Day-2-Day-1、Day0、Day2、Day7、Day9、Day14、Day16、Day21、Day28、Day60 and Day90 post infusion
  Changes in the number of CD56+/ CD3 Anti-PSMA CAR-NK Cell in peripheral blood over time
The pharmacodynamics analysis of Anti-PSMA CAR NK Cell | Baseline to infusion date、Day0、Day1、Day2、Day7、Day8、Day9、Day14、Day15、Day16、Day21、Day28、Day60、Day90、Day120、Day180、Day270 and Day360
  Changes of total prostate specific antigen (tPSA) and free prostate specific antigen (fPSA) in peripheral blood
The proportion of patients with a decrease in PSA levels from baseline | Baseline toDay0、Day1、Day2、Day7、Day8、Day9、Day14、Day15、Day16、Day21、Day28、Day60、Day90、Day120、Day180、Day270 and Day360 post infusion
  PSA response rate
Progression-free survival (PFS) after Anti-PSMA CAR NK Cell infusion | Baseline to 1 year post infusion
  Survival time of patients
Time to clinical progression | Baseline to Day28、Day90、Day180、Day270 and Day360 post infusion
  The time from baseline to the appearance of increased PSA levels or imaging progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, 不限, China